CLINICAL TRIAL: NCT01737255
Title: Magnetic Resonance Imaging Screening In Li Fraumeni Syndrome: An Exploratory Whole Body MRI Study
Brief Title: Magnetic Resonance Imaging Screening in Li Fraumeni Syndrome
Acronym: SIGNIFY
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR3802
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Li-Fraumeni Syndrome
Keywords: Li-Fraumeni Syndrome; Whole Body Magnetic Resonance Imaging; TP53; Psychological Impact
MeSH Terms: conditions — Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TP53 mutation carriers: Carriers of TP53 mutation not known to be low penetrance
  Interventions: Other: Whole body MRI; Other: Psychological questionnaires
- Population controls: Population controls will be sex and aged matched (+/- 5 years) to the TP53 mutation carrier group, with no personal history of cancer and no family history of cancer diagnosed under 50 years
  Interventions: Other: Whole body MRI; Other: Psychological questionnaires

INTERVENTIONS:
Other: Whole body MRI — Individuals will undergo whole body and brain MRI
Other: Psychological questionnaires — All recruits will complete questionnaires at 6 time points to assess psychological impact

SUMMARY:
This study is aimed at exploring the use of whole body MRI for early cancer detection in TP53 mutation carriers and population controls, with the hypothesis that more cancers will be detected in the TP53 mutation carrier group. A secondary end-point will be the number of incidental findings detected and subsequent investigations required. A series of questionnaires will be used to assess the psychological impact of screening on both the study and control group.

ELIGIBILITY:
Inclusion Criteria:

* Carrier of germline TP53 mutation which, in the view of the geneticist, is not known to be low penetrance OR non-related individual with no personal history of malignancy and no first degree relatives diagnosed with malignancy under the age of 50 years
* Please note, TP53 carrier cohort is complete and no longer open to recruitment
* Age between 18 and 60
* Able to give informed consent

Exclusion Criteria:

* Individual with low penetrance TP53 mutation
* Individual with TP53 variant of unknown significance.
* Previous malignancy diagnosed < 5 years ago in TP53 carriers (except non-melanomatous skin cancer or cervical CIS) Previous history of malignancy in non-related controls (except non-melanomatous skin cancer or cervical CIS)
* Current symptoms suggestive of malignancy
* Contraindication to MRI (such as non-MR compatible metal implants) as specified by the standard MR safety checklist
* Claustrophobia
* ECOG performance status >2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The TP53 mutation carriers will be recruited from genetics clinics and through advertising.
  The population controls will be recruited through advertising
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of malignant disease | Within 12 months of MRI scan
  Following MRI scan further investigations may be required to diagnose malignancy

SECONDARY OUTCOMES:
Diagnosis of relevant non-malignant disease | 12 months following MRI scan
  Further investigations may be required following the MRI to characterise such findings.
Diagnosis of non-relevant disease, number and type of investigations required | 12 months following MRI
Psychological impact of MRI screening | 12 months following MRI screening
  Psychological questionnaires to be completed at intervals up till 12 months post scan

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Eeles, PhD, Principal Investigator — Institute of Cancer Research, Surrey, UK
Locations (1):
- Cancer Genetics Unit, Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Steering Committee